CLINICAL TRIAL: NCT06935734
Title: Colonoscopy With a Robotic Endoscope, The CARE I Study
Brief Title: Robotic Colonoscopy Using the Triton 4.0 System in Adults for Screening, Surveillance, and Diagnosis of Lower Gastrointestinal Conditions
Acronym: CARE I
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Neptune Medical (Industry)
Collaborators: KCRI (Other); H-T. Centrum Medyczne Sp. z o.o. sp. k (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CP-000001
Record Dates: First submitted 2025-03-20; First posted 2025-04-20 (Actual); Last update posted 2025-04-20 (Actual); Status verified 2025-04

CONDITIONS: Colonoscopy; Colorectal Cancer Screening; Colorectal Neoplasms; Gastrointestinal Endoscopy
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single Arm (Other): This study is a prospective, single-arm, non-randomized, single site first-in-human study and will be conducted in two phases, where the first phase (A) will serve to evaluate the safety of the Triton 4.0 System to perform screening, surveillance and diagnostic colonoscopies, and the second phase (B) will evaluate the safety and efficacy of the Triton 4.0 System to perform screening, surveillance and diagnostic colonoscopies.
  Interventions: Diagnostic Test: Diagnostic Colonoscopy

INTERVENTIONS:
Diagnostic Test: Diagnostic Colonoscopy — Phase A will serve to evaluate the safety of the Triton 4.0 System to perform screening, surveillance and diagnostic colonoscopies, and Phase B will evaluate the safety and efficacy of the Triton 4.0 System to perform screening, surveillance and diagnostic colonoscopies.

SUMMARY:
This study is a prospective, single-arm, non-randomized, single site first-in-human study and will be conducted in two phases, where Phase A will serve to evaluate the safety of the Triton 4.0 System to perform screening, surveillance and diagnostic colonoscopies, and Phase B will evaluate the safety and efficacy of the Triton 4.0 System to perform screening, surveillance and diagnostic colonoscopies.

ELIGIBILITY:
Inclusion Criteria

1. Age ≥ 22 years
2. Adults indicated for elective screening, surveillance or diagnostic colonoscopy
3. Subject is willing and able to provide written informed consent prior to receiving any non-standard of care Clinical Investigation Plan specific procedures
4. Subject is willing and able to comply with all Clinical Investigation Plan required preparation and follow- up visits -

Exclusion Criteria:

Initial Screening / Pre-Operative:

1. Any medical or physical condition/limitation that would contraindicate a conventional colonoscopy. This assessment will be made by the investigator.
2. Any active implantable medical devices (e.g., pacemakers, defibrillators)
3. Previous failed colonoscopy (except for inadequate bowel preparation)
4. BMI > 45 kg/m2
5. Pregnant participants, women of reproductive potential (pre-menopausal and/or no history of hysterectomy), confirmed by a positive pregnancy test (serum).
6. Surgically altered colonic anatomy
7. History of colorectal cancer, inflammatory bowel disease, polyposis syndrome, hereditary nonpolyposis colorectal cancer (Lynch) syndrome, sclerosing encapsulating peritonitis, active diverticulitis in last 6 months or toxic megacolon
8. Lower gastrointestinal bleeding within 28 days prior to the colonoscopy day
9. Known bleeding tendency such as hemophilia or coagulation factor deficiencies
10. Patient receiving antiplatelet or anticoagulation therapy apart from low-dose aspirin
11. Known colonic stricture
12. Known risk factors for abdominal adhesions such as history of complex abdominal or pelvis surgical procedures, based on investigator assessment
13. Known abdominal wall hernias
14. History of radiotherapy to the abdomen or pelvis
15. History of mesenteric ischemia
16. Known coronary ischemia or cardiovascular stroke within 3 months prior to the colonoscopy procedure
17. Contraindication to the proposed sedation / anesthesia
18. Received any investigational medicine or treatment within 28 days prior to the colonoscopy procedure
19. Received or planning to receive any other endoscopic procedure within 4 weeks prior and 2 weeks after the colonoscopy procedure
20. Participation in any concurrent clinical trial that may impact the results of this study

    Intra-Operative Exclusion Criteria:
21. Inadequate Bowel Preparation, Boston Bowel Prep Scale Score (after cleansing) < 2 in any section
22. Failed conventional colonoscopy or polypectomy/biopsy performed during the conventional colonoscopy procedure in Phase A
23. Any presenting condition discovered intraoperatively that in the opinion of the investigator would make participating in this study not in the participant's/patient's best interest. For example, presence of a stricture or tight sigmoid that would make passing an overtube risky for the patient
24. Any condition, in the opinion of the Investigator, that is unstable and could jeopardize the safety of the subject and their compliance in the study

Min Age: 22 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-04-14 (Estimated); Primary Completion 2025-06-06 (Estimated); Study Completion 2025-07-31 (Estimated)

PRIMARY OUTCOMES:
Safety Endpoint - Incidence of Major Adverse Events Within 48 Hours | 48 hours
  Absence of Major Adverse Events (MAEs) within 48 hours of the procedure. MAEs are defined as any of the following:
  1. Device-related death within 48 hours
  2. Perforation within 48 hours
  3. Intraprocedural bleeding preventing completion of the procedure
  4. Delayed bleeding within 48 hours accompanied by pre-defined symptoms and confirmed by a hemoglobin drop of >2 g, leading to admission to the hospital, prolongation of hospital stay, or another procedure requiring sedation/anesthesia.
  Unit of Measure: Number of participants with at least one Major Adverse Event
Efficacy Endpoint - Successful Completion of Colonoscopy | During procedure
  Completion of colonoscopy defined by both: (a) successful cecal intubation (clinically acceptable access and visualization of the cecum), and (b) successful withdrawal (clinically acceptable diagnostic and therapeutic access of the entire colon tract).

SECONDARY OUTCOMES:
Time to Cecum | During procedure
  Time from scope insertion to successful cecal intubation. Unit of Measure: Minutes
Need for Repositioning | During procedure
  Number of times a participant was repositioned to facilitate scope advancement. Unit of Measure: Number of repositioning events
Polypectomy Success | During procedure
  If applicable, indicates whether at least one polyp was successfully removed using standard polypectomy tools during the procedure. This outcome is evaluated per participant and applies only to Phase B (robotic procedures).
  Unit of Measure: Categorical - Yes / No / Partial (i.e., at least one polyp removed, but not all targeted polyps).
NASA Task Load Index (NASA-TLX) | Post-procedure
  Physician's subjective workload assessment using the NASA Task Load Index (NASA-TLX), a validated tool consisting of six subscales: Mental Demand, Physical Demand, Temporal Demand, Performance, Effort, and Frustration. Each subscale is scored from 0 to 100 in increments of 5. Higher scores indicate greater perceived workload.
  Unit of Measure: Composite score (0-100)
Mucosal Injury Score | During procedure
  Mucosal injury graded using a 5-point ordinal scale based on injury severity: 1 = Erythema/ Bruising, 2 = Mucosal break <5mm in length, 3 = Mucosal break >5mm in length, 4 = Mucosal Injury (non-full thickness), 5 = Full thickness injury. Outcome is reported per subject. Only applicable to Phase B (robotic procedures).
  Unit of Measure: Score (1-5); higher scores indicate more severe injury
Delayed Bleeding (14 Days) | 14 days
  Number of participants with delayed bleeding within 14 days confirmed by pre-determined symptoms and hemoglobin drop of >2 g/dL.
  Unit of Measure: Number of participants
Delayed Perforation (14 Days) | 14 days
  Number of participants with delayed perforation identified within 14 days post-procedure.
  Unit of Measure: Number of participants
Adenoma Detection Rate (ADR) | During procedure
  Proportion of participants in whom at least one adenomatous polyp is detected during the robotic colonoscopy procedure. Applicable to Phase B (robotic procedures) only.
  Unit of Measure: Percentage of participants with ≥1 adenoma detected

CONTACTS AND LOCATIONS:
Overall Officials: Marcin Romanczyk, Principal Investigator — H-T Centrum Medyczne; Jason Samarasena, MD, Principal Investigator — University of California, Irvine; Tomasz Romanczyk, Principal Investigator — H-T Centrum Medyczne